CLINICAL TRIAL: NCT03464851
Title: Evaluation of a Novel Technique to Diagnose Carotid Artery Stenosis
Status: Terminated | Type: Observational
Why Stopped: Low enrollment due to inclusion/exclusion criteria
Sponsor: The Cleveland Clinic (Other)
Collaborators: CVR Global, Inc. (Industry)
Responsible Party: Principal Investigator, Imad Bagh, M. D., Principal Investigator, The Cleveland Clinic
Other Study IDs: IRB 18-126
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stenosis; plaque; carotid duplex; ultrasound; fibromsucular dysplasia; carotid atherosclerosis
MeSH Terms: conditions — Carotid Stenosis; Plaque, Amyloid; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unknown/Normal/Mild Disease: No prior carotid duplex study or known normal or mild disease in the ICAs (PSV <= 125 cm/sec)
  Interventions: Diagnostic Test: Carotid Stenotic Scan (CSS)
- Known moderate or severe ICA Stenosis (PSV>125 cm/sec)
  Interventions: Diagnostic Test: Carotid Stenotic Scan (CSS)
- Known ICA Fibromuscular Dysplasia
  Interventions: Diagnostic Test: Carotid Stenotic Scan (CSS)

INTERVENTIONS:
Diagnostic Test: Carotid Stenotic Scan (CSS) — Placement of the CSS instrument on the carotid arteries to measure degree of stenosis
  of the carotid artery. The CSS scan takes about 1-2 minutes to gather data for real-time analysis by the processor on the device cart.

SUMMARY:
The purpose of this study is to determine the accuracy of a new non-invasive device, the Carotid Stenotic Scan (CSS), to check for stenosis of the internal carotid artery (ICA) as compared to a carotid ultrasound study.

DETAILED DESCRIPTION:
Currently, carotid duplex ultrasound is used for screening for ICA stenosis and must be performed by a trained and certified vascular technologist using advanced duplex imaging equipment and with subsequent interpretation by a trained physician. It would be of value to develop an accurate, reliable, low-cost, and easily accessible tool to screen for extra-cranial ICA disease in an office based setting. However, such a tool would require novel technology that allows for quick, accurate, reproducible, and safe evaluation.

This study will evaluate a new technology called the Carotid Stenotic Scan (CSS) developed by CVR Global. The CSS instrument uses principles of cardiovascular resonance to detect low frequency pressure fluctuations associated with flow disturbances in areas of significant arterial narrowing.

Subjects will undergo a clinically ordered clinical carotid duplex ultrasound as part of standard of care. Subjects will have a noninvasive CSS assessment before or after the carotid duplex ultrasound.

Within 3 months following the date of the initial study visit, the electronic medical record will be queried for any interval correlative imaging studies (CTA, MRA, or angiography) and reports performed up to 1 month prior and 3 months after the duplex examination date. Report of findings will be documented (i.e., % ICA stenosis by CTA/MRA).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients age > 18 years sent to the vascular laboratory for carotid duplex examination for initial carotid ultrasound study or for follow-up of known carotid disease.
* Enrolled patients will include at least 100 subjects with at least moderate known stenosis (50-69% or greater, PSV > 125 cm/sec) or occlusion of one or both ICAs
* Up to 25 patients with known fibromuscular dysplasia (FMD) of the internal carotid arteries.

Exclusion Criteria:

* Age < 18 years.
* Hospitalized inpatients.
* Inability to provide informed consent.
* Prior history of carotid endarterectomy or carotid artery stent.
* Prior neck surgery
* Known prosthetic heart valve, known critical aortic stenosis, or study indication "preop" open heart or aortic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consistent of adult patients (> 18 years) presenting to the Cleveland Clinic Non-Invasive Vascular Laboratory for a scheduled carotid duplex ultrasound to evaluate for carotid artery disease or in follow-up of known ICA stenosis.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Comparison of CSS readings to conventional carotid artery duplex ultrasound | Baseline
  Primary analysis % agreement CSS and carotid duplex ultrasound (SRUCC interpretation) for ICA stenosis

SECONDARY OUTCOMES:
Reproducibility of the CSS measurement | Baseline
  Each CSS measurement will be repeated and the Intraclass Correlation Coefficient (ICC) will be calculated. The ICC in an index of the reliability of measurements from the same operator

CONTACTS AND LOCATIONS:
Overall Officials: Imad Bagh, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT03464851/Prot_000.pdf
  • Informed Consent Form (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03464851/ICF_001.pdf